CLINICAL TRIAL: NCT02359149
Title: Intravitreal Injections by Nurses or Physicians: a Randomized Controlled Trial Comparing Efficacy, Patient Satisfaction and Health Economy
Brief Title: Intravitreal Injections by Nurses and Physicians Compared
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/1719
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Eye Diseases
Keywords: Intravitreal injections; Nurses; Physicians
MeSH Terms: conditions — Eye Diseases | interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse (Experimental): intravitreal injections with anti-VEGF agents given by a nurse
  Interventions: Procedure: intravitreal injections given by a nurse; Procedure: Intravitreal injections; Drug: Anti-VEGF agents
- physician (Active Comparator): intravitreal injections with anti-VEGF agents given by a physician
  Interventions: Procedure: intravitreal injections given by a physician; Procedure: Intravitreal injections; Drug: Anti-VEGF agents

INTERVENTIONS:
Procedure: intravitreal injections given by a nurse
  Arms: nurse
Procedure: intravitreal injections given by a physician
  Arms: physician
Procedure: Intravitreal injections
Drug: Anti-VEGF agents
  Other Names: anti vasculer endothelial growth factor

SUMMARY:
Anti-VEGF agents are given for a variety of previously untreatable eye diseases. The last years indications for their use and consequently the number of patients needing treatment, have been increasing. Most patients require multiple injections. This has resulted in many eye departments administering thousands of injections per year, also at St Olavs University Hospital Trondheim. To cope with this increase in workload, it would be helpful if injections would be given not only by the physicians but also by the nurses. This study's objective is to compare efficiency, patient satisfaction and cost per patient of injections given by nurses and physicians.

ELIGIBILITY:
Inclusion Criteria:

* referred to the eye clinic for treatment of age related macular degeneration, diabetes retinopathy or retinal vein occlusion with anti-vascular endothelium growth factor
* Ability to provide written informed consent
* ability to comply with study assessments for the full duration of the study

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
change in visual acuity | 1 year
  Mean change in visual acuity from baseline to 12 months, tested on ETDRS letter chart

SECONDARY OUTCOMES:
incidence of ocular adverse events | from baseline to 12 months
patient satisfaction | 12 months
  questionnaire after the first treatment will be compared with questionnaire after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marit Fagerli, md, Study Director — St. Olavs University Hospital
Locations (1):
- St Olavs Hospital, Department of Ophthalmology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austeng D, Morken TS, Bolme S, Follestad T, Halsteinli V. Nurse-administered intravitreal injections of anti-VEGF: study protocol for noninferiority randomized controlled trial of safety, cost and patient satisfaction. BMC Ophthalmol. 2016 Oct 1;16(1):169. doi: 10.1186/s12886-016-0348-4. PMID 27716253
- [Result] Bolme S, Morken TS, Follestad T, Sorensen TL, Austeng D. Task shifting of intraocular injections from physicians to nurses: a randomized single-masked noninferiority study. Acta Ophthalmol. 2020 Mar;98(2):139-144. doi: 10.1111/aos.14184. Epub 2019 Jul 3. PMID 31267688
- [Derived] Bolme S, Austeng D, Morken TS, Follestad T, Halsteinli V. Cost consequences of task-shifting intravitreal injections from physicians to nurses in a tertiary hospital in Norway. BMC Health Serv Res. 2023 Mar 8;23(1):229. doi: 10.1186/s12913-023-09186-0. PMID 36890535